CLINICAL TRIAL: NCT05018455
Title: The Effectiveness of Remote Fall Prevention Program vs. Face-to-Face in Low-medium Risk Elderly- A Cross Over Randomized Controlled Trial
Brief Title: The Effectiveness of Remote Fall Prevention Program vs. Face-to-Face
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Remote fall prevention
Record Dates: First submitted 2021-08-16; First posted 2021-08-24 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2022-08

CONDITIONS: Fall
Keywords: Telehealth, fall prevention, home dwelling elderly, Otago

STUDY DESIGN:
Intervention Model Description: The intervention program will include Otago- based fall prevention training face-to-face or remote. Each subject will receive the two types of interventions in sequence, with a cooling-off period between them. The intervention program in this study will last 6 months, however, the intervention arm will be swapped after 3 months.
Who Masked: Outcomes Assessor
Masking Description: Functional and balance tests will be performed by a skilled physiotherapist, blind to the participant's group affiliation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fall prevention intervention program conducted through telehealth (Experimental): The training program is based on the principles of the Otago program, designed specifically to prevent falls. It consists set of leg muscle strengthening and balance retraining exercises progressing in difficulty, and a walking plan. The training will be delivered to a group of 10 participants. Each participant will practice from home, using a zoom system. The duration of each training will be one hour, the frequency of training will be twice a week for three months.
  Interventions: Other: Fall prevention program training based on Otago principles
- Similar fall prevention intervention program conducted through face to face group training (Active Comparator): The training program is based on the principles of the Otago program, designed specifically to prevent falls. It consists set of leg muscle strengthening and balance retraining exercises progressing in difficulty, and a walking plan. The training will be delivered to a group of 10 participants. The training sessions will be delivered at the local community center, twice a week for one hour for three months.
  Interventions: Other: Fall prevention program training based on Otago principles

INTERVENTIONS:
Other: Fall prevention program training based on Otago principles — balance and strength exercises

SUMMARY:
Falls are a serious problem in the elderly leading to injuries, morbidity, and consequently a heavy impact on the individual suffering, and society at large.

This study aims to investigate the effectiveness of a remote fall prevention program in comparison with a similar face-to-face program. This study design is a randomized control trial (RCT) with a cross-over in group allocation. The population will include 106 home-dwelling elderly, aged 65 years or more, with low to moderate risk of fall. Participants will be randomized to start intervention in the remote or face-to-face group. Training will be twice weekly for 3 months, after which there will be two weeks of washout, followed by a cross-over between groups. Outcome measures will include fall rate over a year (primary measure), balance, functional testing, subjective measures of fear of falls, quality of life, satisfaction from intervention, adherence, and compliance.

DETAILED DESCRIPTION:
The aim of the proposed study is to investigate the effectiveness of a remote fall prevention training program. The proposed intervention program includes an Otago-based fall prevention training program to improve lower extremity strength, balance, and walking, directed by physical therapists, over 6 months. The remote group will train at home, using video communication software, while the face-to-face group will train at a local community center.

The proposed study will be designed as a randomized control trial (RCT) with a cross-over design. The population will include 106 home-dwelling elderly, aged 65 years or more, walking independently, that will be identified at low to moderate risk of fall. Candidates with unbalanced systemic disease or disorders, cognitive and physical Impairments that will prevent participation in the program, will not be included. A full description of the inclusion and exclusion criteria is provided below in the Eligibility section.

Participants will be randomized into two groups that will receive similar Otago-based fall prevention group training, either remotely or face-to-face.

The training sessions: The training starts with five minutes of gentle warm-up with the same five flexibility exercises, followed by structured lower limb muscles strengthening, balance exercises, and instruction for independent walking for up to 30 minutes at least twice a week. The training will be delivered to groups of ten participants. The duration of each session will be one hour, twice a week for three months. After three months of training, there will be a two weeks break, serving as a washout period, after which the groups will switch, for another three months. At the end of the intervention period (6.5 months), each participant will be trained by both remote and face-to-face programs. Assessments will be conducted at 4-time points: baseline, 3 months after completion of the first-ordered training, 6.5 months after completion of both trainings, and 12 months follow up.

The primary outcome measure is the number of falls during a year. secondary outcome measures include Objective measures as balance, Walking speed, lower extremities functional strength, adherence, and compliance to the training program. The subjective outcome measure will include participant Satisfaction from the program, Fear of falls, and Quality of life. More details regarding outcome measures are provided below in the outcome measure section.

Statistical analysis: The equivalence test will be used to examine if the remote fall prevention training is as good as the face-to-face. In order to check if there is a period-treatment effect on the objective outcome measures we will employ a mixed-model repeated-measures analysis of variance (ANOVA): 4-time points (baseline, 3 months, 6 months, 12 months follow up) X 2 interventions (remote vs. face-to-face), counting for the fact that subjects are nested in sequence. When interaction will be significant simple mean analysis will be used to reveal a significant source. Studentized Maximum Modulus (SMM) post-hoc adjustment method will be used to reveal significance between pairs of periods.

If this study will manage to show remote fall prevention is feasible, safe, and effective, it will promote a solution in one of the most serious health problems in the elderly, in one of the most challenging eras for the elderly, when remote healthcare is vital.

ELIGIBILITY:
Inclusion Criteria:

* home-dwelling elderly, aged 65 years or more
* Identified to be at low to moderate risk of falling

Risk of falling will be assessed according to a combination of subjective and objective evaluation. Subjective questions from the STEADI (stopping elderly accidents death, and injuries), an algorithm for fall risk screening, assessment, and intervention, developed by the American Center for Disease Control and Prevention, relate to (1) Feels unsteady when standing/walking, (2) Worries about falling, and (3) Has fallen no more than 3 times in the past year.

An additional inclusion criterion is scoring 21 or more in the Mini-Best test (a balance test).

Exclusion Criteria:

* Subjects suffering from severe musculoskeletal pain or disorders that will limit completion of the assessment procedure such as pain limiting weight-bearing for no longer than a few minutes
* Unstable cardiovascular/pulmonary disease
* Unbalanced diabetes
* Neurological diseases such as stroke, Parkinson's, or multiple sclerosis
* Use of a walking aid (except for a cane)
* visual or hearing impairment that will not allow the use of technology for remote practice
* A score lower than 21/30 on the Montreal Cognitive Assessment score (MoCA),
* High risk of falling on the balance test (Mini-BESTest ≤ 20)

Comment: exclusion criteria will be based on self-report and completed at the initial baseline assessment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Number of falls during the study period | Falls will be monitored for one year
  Subjects will self-report falls weekly in a personal fall diary. This will be supported by a telephone call from one of the investigators once a month.

SECONDARY OUTCOMES:
Mini Balance Evaluation Systems Tests | Change from baseline at 3, 6 and 12 months
  Mini Balance Evaluation Systems Tests (Mini-BESTest) is a clinical balance assessment tool. This test includes 14 items, each scored from 0 (severe balance impairment) to 2 (no balance impairment). The maximal possible score is 28 points. Higher scores indicate better balance performance. A score of 20 points or below indicates a high fall risk.
Time-Up and Go Test | Change from baseline at 3, 6 and 12 months
  The Timed Up and Go Test (TUG) assesses mobility, balance, and fall risk in older adults. The test measures the time required for a subject to stand up from sitting on a chair, walk for 3 meters, turn, walk back, and sit down. A score of 12 seconds or more indicates risk of falling in community dwelling adults.
Berg Balance Scale | Change from baseline at 3, 6 and 12 months
  The Berg Balance Scale (BBS) is a 14- item objective measure that assesses static and dynamic balance, and fall risk in adults. Each item is scored from 0 (unable to perform) to 4 (normal performance). The maximal possible score is 56 points. Any score from 0 to 36 indicate 100% fall risk for older adults. The Berg Balance Scale (BBS) is widely used in clinical practice to predict falls in the older adults. lately, due to ceiling effect, the use of BBS as a single measure to accurately predict future falls seems to be insufficient.
Four Stage Balance Test | Change from baseline at 3, 6 and 12 months
  The 4-Stage Balance Test assess static balance at four standing positions, that get progressively harder to maintain. The person is asked to hold a position for 10 seconds without moving his feet or supporting. An older adult, who cannot hold the tandem stand, which is the forth position, for at least 10 seconds, is at increased risk of falling.
Walking speed | Change from baseline at 3, 6 and 12 months
  Walking speed will be measured using the 4-Meter Walk Test in seconds. Walking speed lower than 1.0 seconds/meter is considered a strong predictor of falls in the elderly population living in the community.
Lower extremities functional strength | Change from baseline at 3, 6 and 12 months
  Functional strength of the lower limbs will be measured by the 30-second Sit to Stand Test. This is also used for fall prediction. A result lower than expected by age and sex indicates a risk of falls
Attendance | Will be monitored and record in any session time, for 6 months
  Attendance to the program will be recorded each class by the physiotherapist who will conduct the training. Total attendance will be defined as the number/percentage of classes attended out of the total number of sessions conducted, for example attending 75 sessions out of 100 will be calculated as total attendance of 75%.
Completion (retention) | Will be monitored and record in any session time, for 6 months
  Completion of the full period of the program- 6 months, will be recorded for each participant, and will reflect retention. Non-completion will be recorded for the participants who will withdrawal from the program before the end of the program, and will not complete the 6 months, end of program, assessment.
Satisfaction from program | Twice- after each program session (after 3 and 6 months).
  Participant satisfaction will be assessed using a satisfaction rating scale of 0-10, with a score of 0 indicating complete dissatisfaction and a score of 10 maximum satisfaction.
Fear of falls | Change from baseline at 3, 6 and 12 months
  Fear of falls will be assessed using the Modified Falls Efficacy Scale (MFES) questionnaire, which is one of the most common and reliable research tools in fall research. In this questionnaire, the subject rates his confidence in performing 10 daily tasks
12-Item Short Form Survey (SF-12) Quality of life questionnaire | Change from baseline at 3, 6 and 12 months
  Quality of life will be assessed using the SF-12 questionnaire. This questionnaire assesses the perception of quality of life through 12 questions that relate to the subject's views about his state of health and ability to perform various actions and functions. The use of this questionnaire is common in fall studies.

CONTACTS AND LOCATIONS:
Overall Officials: Hilla Sarig Bahat, PT PhD, Principal Investigator — Department of Physical Therapy, University of Haifa
Locations (2):
- Israel (2):
  - The Faculty of Social Welfare and Health Science, Haifa University, Haifa
  - Gold club Kfar vradim, Kfar Vradim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sherrington C, Fairhall NJ, Wallbank GK, Tiedemann A, Michaleff ZA, Howard K, Clemson L, Hopewell S, Lamb SE. Exercise for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2019 Jan 31;1(1):CD012424. doi: 10.1002/14651858.CD012424.pub2. PMID 30703272
- [Background] Kyrdalen IL, Moen K, Roysland AS, Helbostad JL. The Otago Exercise Program performed as group training versus home training in fall-prone older people: a randomized controlled Trial. Physiother Res Int. 2014 Jun;19(2):108-16. doi: 10.1002/pri.1571. Epub 2013 Dec 11. PMID 24339273
- [Background] Bernocchi P, Giordano A, Pintavalle G, Galli T, Ballini Spoglia E, Baratti D, Scalvini S. Feasibility and Clinical Efficacy of a Multidisciplinary Home-Telehealth Program to Prevent Falls in Older Adults: A Randomized Controlled Trial. J Am Med Dir Assoc. 2019 Mar;20(3):340-346. doi: 10.1016/j.jamda.2018.09.003. Epub 2018 Oct 23. PMID 30366759
- [Derived] Toledano-Shubi A, Livne D, Hel-Or H, Bahat HS. Remote fall prevention training for community-dwelling older adults: comparison with face-to-face and effect of delivery sequence-A randomized controlled trial. Geriatr Nurs. 2026 Jan 21;69:103817. doi: 10.1016/j.gerinurse.2026.103817. Online ahead of print. PMID 41570620
- See also: Centers for Disease Control and Prevention. STEADI- Older adult fall prevention — https://www.cdc.gov/steadi/index.html
- See also: Otago Exercise Programme to prevent falls in older adults — https://www.livestronger.org.nz/assets/Uploads/acc1162-otago-exercise-manual.pdf